CLINICAL TRIAL: NCT06516705
Title: The Relationship Between Knowledge, Self-care Behaviors, Fear, Social Support and Quality of Life in Patients With Type 2 Diabetes, and the Effectiveness of Multimedia Education on Hypoglycemic Management.
Brief Title: The Effectiveness of Multimedia Education on Hypoglycemic Management.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KMUHIRB-E(II)-20180100
Record Dates: First submitted 2024-07-09; First posted 2024-07-24 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-07

CONDITIONS: Type2diabetes; Hypoglycemia
Keywords: multimedia education; hypoglycemia; knowledge; self-care behavior; the recurrence rate of hypoglycemic events
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Participants in the experimental group receiving multimedia hypoglycemia education and participants in the contrast group receiving conventional hypoglycemia education.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimedia hypoglycemia health education (Experimental): The multimedia educational content included an introduction to blood glucose, symptoms and management of hypoglycemia (the 15-rule), prevention of hypoglycemia (diet and exercise), and medication therapy.
  Interventions: Behavioral: Hypoglycemia education
- Conventional hypoglycemia education (Active Comparator): The verbal educational content provided by the health educators included an introduction to blood glucose, symptoms and management of hypoglycemia (the 15-rule), prevention of hypoglycemia (diet and exercise), and medication therapy.
  Interventions: Behavioral: Hypoglycemia education

INTERVENTIONS:
Behavioral: Hypoglycemia education — Hypoglycemia education : incleded introduction to blood glucose, hypoglycemia symptoms and treatment (15-15 rule), prevention of hypoglycemia (diet and exercise), and medication treatment.

SUMMARY:
The first phase of the research was to develop tools, including scales and multimedia, and the second phase was to carry out multimedia hypoglycemia education intervention measures. An experimental randomized controlled trial with a repeated measures design was conducted in second phase. Participants in the experimental group receiving multimedia hypoglycemia education and participants in the contrast group receiving conventional hypoglycemia education. Structural questionnaires were used for data collection. The study was to investigate the effectiveness of multimedia hypoglycemia education compared to conventional hypoglycemia education on knowledge, self-care behavior, fear of hypoglycemia, social support, quality of life, nursing hours, education satisfaction, and the recurrence rate of hypoglycemic events among patients with type 2 diabetes.

DETAILED DESCRIPTION:
In the first phase, we created multimedia educational content on hypoglycemia and recruited 300 type 2 diabetes patients who had experienced hypoglycemic events from a medical center and a primary care clinic in southern Taiwan. The participants completed consent forms and questionnaires, and we conducted statistical analyses to develop and evaluate knowledge and behavior assessment tools. We obtained consent from 83 participants to enter the second phase, where they received hypoglycemia education and were then randomly assigned by computer to either the experimental group or the contrast group.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes and blood glucose levels below 70 mg/dL

Exclusion Criteria:

* patients with cognitive impairment, those who are unable to perform activities of daily living and those with severe or unstable medical conditions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: T1( Before Hypoglycemia Education)
Arm/Group | Multimedia Hypoglycemia Health Education | Conventional Hypoglycemia Education
Started | 42 | 41
Completed | 41 | 41
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: T2( After Hypoglycemia Education)
Arm/Group | Multimedia Hypoglycemia Health Education | Conventional Hypoglycemia Education
Started | 41 | 41
Completed | 41 | 41
Not Completed | 0 | 0
Period: T3 ( 3 Month After Education)
Arm/Group | Multimedia Hypoglycemia Health Education | Conventional Hypoglycemia Education
Started | 41 | 41
Completed | 37 | 35
Not Completed | 4 | 6
Not completed — No follow-up clinic visits | 3 | 3
Not completed — covid-19 | 1 | 2
Not completed — Refused to respond | 0 | 1
Period: T4 ( 6 Month After Education)
Arm/Group | Multimedia Hypoglycemia Health Education | Conventional Hypoglycemia Education
Started | 41 | 41
Completed | 35 | 35
Not Completed | 6 | 6
Not completed — No follow-up clinic visits | 3 | 3
Not completed — covid-19 | 3 | 2
Not completed — Refused to respond | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multimedia Hypoglycemia Health Education | Conventional Hypoglycemia Education | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 30 | 32 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (7.2) | 69.7 (5.6) | 69.9 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 37
  Male | 25 | 20 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 41 | 41 | 82
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 41 | 41 | 82

OUTCOME MEASURES:

1. Primary Outcome: The Score of Hypoglycemia Knowledge
Description: Hypoglycemia management knowledge scale to collect the score in Knowledge. The scale consists of eight true/false questions, with scores ranging from 0 to 8 points. Higher scores indicate a higher level of knowledge about hypoglycemia in patients.
Time Frame: Through study completion, an average of 6 months after education.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Multimedia Hypoglycemia Health Education | Conventional Hypoglycemia Education
Number analyzed (Participants) | 41 | 41
score on a scale | 5.8 (0.2) | 4.8 (0.2)

2. Primary Outcome: The Score of Hypoglycemia Self-care Behavior
Description: Hypoglycemia self-care behavior scale to collect the score in Behavior. The scale comprises 10 items, each rated on a 5-point Likert scale, with total scores ranging from 10 to 50. Higher scores indicate better self-care behaviors in managing hypoglycemia.
Time Frame: Through study completion, an average of 6 months after education.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Multimedia Hypoglycemia Health Education | Conventional Hypoglycemia Education
Number analyzed (Participants) | 41 | 41
score on a scale | 31.2 (0.8) | 28.6 (0.9)

3. Primary Outcome: Nursing Time
Description: Form Recorded for Health Education Time
Time Frame: Through study completion, an average of 6 months after education.
Measure: Mean (Standard Deviation); unit: minute
Arm/Group | Multimedia Hypoglycemia Health Education | Conventional Hypoglycemia Education
Number analyzed (Participants) | 41 | 41
minute | 9.4 (2.4) | 14.8 (7.0)

4. Primary Outcome: The Score of Education Satisfaction
Description: Education satisfaction scale to collect the score in education satisfaction. Items were rated on a 5-point Likert scale, with a score range of 1 to 5 points, for a total score range of 5 to 25 points.
Time Frame: Through study completion, an average of 6 months after education.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Multimedia Hypoglycemia Health Education | Conventional Hypoglycemia Education
Number analyzed (Participants) | 41 | 41
score on a scale | 22.6 (4.5) | 17.1 (4.3)

5. Primary Outcome: The Recurrence Rate of Hypoglycemic Events
Description: Questionnaire to assess the rate of hypoglycemic events.
Time Frame: Through study completion, an average of 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Multimedia Hypoglycemia Health Education | Conventional Hypoglycemia Education
Number analyzed (Participants) | 41 | 41
Participants | 16 | 19

6. Secondary Outcome: The Score of Fear of Hypoglycemia
Description: Hypoglycemia fear scale to collect the score in fear of hypoglycemia. This scale consists of 13 items, rated on a 5-point Likert scale with a score range of 0 to 52 points. Higher scores indicate a greater degree of fear of hypoglycemia among patients.
Time Frame: Through study completion, an average of 6 months after education.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Multimedia Hypoglycemia Health Education | Conventional Hypoglycemia Education
Number analyzed (Participants) | 41 | 41
score on a scale | 7.0 (0.8) | 5.1 (0.7)

7. Secondary Outcome: The Score of Social Support
Description: Social support scale to collect the score in social support. The scale consists of 13 items, rated on a 5-point Likert scale with a score range of 0 to 52 points. Higher scores indicate higher levels of social support.
Time Frame: Through study completion, an average of 6 months after education.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Multimedia Hypoglycemia Health Education | Conventional Hypoglycemia Education
Number analyzed (Participants) | 41 | 41
score on a scale | 23.0 (1.6) | 21.8 (1.4)

8. Secondary Outcome: The Score of Quality of Life
Description: Quality of life scale to collect the score in quality of life. The scale consists of 28 items, each rated on a 5-point Likert scale, with scores for each domain converted to a total range of 16 to 80 points.
Time Frame: Through study completion, an average of 6 months after education.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Multimedia Hypoglycemia Health Education | Conventional Hypoglycemia Education
Number analyzed (Participants) | 41 | 41
score on a scale | 52.3 (0.8) | 51.5 (0.8)

ADVERSE EVENTS:
Time Frame: The time before education, the time after education, 3 month after education and 6 month after education.
Arm/Group | Multimedia Hypoglycemia Health Education | Conventional Hypoglycemia Education
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT06516705/Prot_SAP_000.pdf